CLINICAL TRIAL: NCT02637440
Title: Multi Centre Open Label Randomised Controlled Parallel-group Three Arm Trial To Compare The Use Of Fractional Flow Reserve (FFR) Guided and Angiographically Guided Revascularization To The Treatment Of Infarct Related Artery Only In Patients With STEMI And Multivessel Disease
Brief Title: The Use Of FFR Guided PCI Versus Complete Revascularization and Treatment Of Infarct Related Artery Only In Patients With STEMI
Acronym: FAIO
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Limerick (Other)
Responsible Party: Principal Investigator, A Abdullah, Dr., University of Limerick
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FA 2015
Record Dates: First submitted 2015-12-17; First posted 2015-12-22 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-12

CONDITIONS: Multivessel Coronary Artery Disease; STEMI; FFR Guided PCI
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Conservative (No Intervention): After the index primary PCI. The control group will receive best medical therapy and regular follow up and only PCI for recurrent angina with evidence of inducible ischaemia.
- FFR guided (Active Comparator): FFR group will undergo FFR at 4 weeks of the index primary PCI as OPD. If FFR is less than 0.8, then PCI will be performed
  Interventions: Procedure: FFR guided PCI
- angiogram guided (Active Comparator): The group will undergo PCI for all significant lesions more than 50
  Interventions: Procedure: Angio guided PCI

INTERVENTIONS:
Procedure: FFR guided PCI — Patients undergo Fractional Flow measurement (FFR) followed by PCI, if the FFR is less than 0.8
  Arms: FFR guided
Procedure: Angio guided PCI — Patients receive PCI without FFR measurement
  Arms: angiogram guided

SUMMARY:
In patients with ST elevation myocardial infarction (STEMI) the treatment goal is revascularization of the occluded artery with the use of primary percutaneous coronary intervention (PCI). There is a large subset of patients with STEMI who also have significant disease in arteries other than the site of occlusion, and away from the culprit artery. It is estimated that up to 50% have disease of more than 50% in the non-culprit arteries.

The evidence on how to treat those patients with multi vessel disease is conflicting. Earlier large-scale studies and registries have suggested early and complete revascularization is of no benefit or even harmful. More recent studies have showed the opposite of that. The CVLPRIT study showed that early complete revascularization or preventive PCI reduced primary endpoint of a composite of all cause mortality, myocardial infarction and need for repeat revascularization. The benefit was mainly due to reduced repeat revascularization in the more intensive intervention group. The PRAMI study showed very similar results as well.

The use of Fractional flow Reserve (FFR) in deciding complete revascularization has also showed conflicting results so far. A previous trial showed that FFR guided intervention post STEMI increased MACE. This was conflicted with more recent study, which showed FFR guided complete revascularization improved outcome when compared with more conservative treatment of ischaemia driven intervention.

In this study, the investigators are going to assess the issue of staged revascularization guided by FFR or by angiogram, compared to the standard treatment of ischaemia driven revascularization

DETAILED DESCRIPTION:
To compare the clinical outcomes measured by composite of mortality, myocardial infarction and repeat revascularization by using FFR guided and angiographically guided revascularization to the standard strategy of ischaemia driven revascularization.

Participants will be allocated to three arms, first conservative group of ischaemia guided PCI, second FFR guided PCI and third angiogram guided PCI where patients where patients with more than 50% lesion will undergo revascularization.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with STEMI and multi-vessel disease on initial angiogram.
2. Above 18 years of age
3. Able to give consent

Exclusion Criteria:

1. Patients with indication for CABG
2. Left main stem lesion of >50%
3. Cardiogenic shock
4. Intractable angina during hospital admission
5. Patients with limited life expectancy
6. Patients with severe chronic kidney disease
7. Patients with contraindication to dual antiplatelet therapy
8. Patients with very complex lesions that deemed not favourable for PCI
9. Pregnancy or childbearing age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Estimated)
Dates: Start 2015-12; Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Composite of cardiovascular death, myocardial infarction and / or revascularization | 1 year

SECONDARY OUTCOMES:
Cardiovascular morality | 1 year
Myocardial infarction | 1 year
Revascularization | 1 year
  Revascularization procedure because of symptoms and evidence of ischaemia
stroke | 1 year
Heart failure | 1 year
  documented episode of presentation with symptoms consistent with heart failure and evidence from echocardiogram or laboratory test consistent with the diagnosis of heart failure
Costs | 1 year
  total procedural costs, hospital stay costs, medications costs.

OTHER OUTCOMES:
Bleeding | 1 year
  any major bleeding (TIMI 3)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Kiernan, MD, Principal Investigator — University Hospital of Limerick
Locations (2):
- Ireland (2):
  - Galway University Hospital, Galway, Galway
  - University Hospital Limerick, Limerick, Limerick

REFERENCES:
- [Background] Gershlick AH, Khan JN, Kelly DJ, Greenwood JP, Sasikaran T, Curzen N, Blackman DJ, Dalby M, Fairbrother KL, Banya W, Wang D, Flather M, Hetherington SL, Kelion AD, Talwar S, Gunning M, Hall R, Swanton H, McCann GP. Randomized trial of complete versus lesion-only revascularization in patients undergoing primary percutaneous coronary intervention for STEMI and multivessel disease: the CvLPRIT trial. J Am Coll Cardiol. 2015 Mar 17;65(10):963-72. doi: 10.1016/j.jacc.2014.12.038. PMID 25766941
- [Result] Levine GN, Bates ER, Blankenship JC, Bailey SR, Bittl JA, Cercek B, Chambers CE, Ellis SG, Guyton RA, Hollenberg SM, Khot UN, Lange RA, Mauri L, Mehran R, Moussa ID, Mukherjee D, Ting HH, O'Gara PT, Kushner FG, Ascheim DD, Brindis RG, Casey DE Jr, Chung MK, de Lemos JA, Diercks DB, Fang JC, Franklin BA, Granger CB, Krumholz HM, Linderbaum JA, Morrow DA, Newby LK, Ornato JP, Ou N, Radford MJ, Tamis-Holland JE, Tommaso CL, Tracy CM, Woo YJ, Zhao DX. 2015 ACC/AHA/SCAI Focused Update on Primary Percutaneous Coronary Intervention for Patients With ST-Elevation Myocardial Infarction: An Update of the 2011 ACCF/AHA/SCAI Guideline for Percutaneous Coronary Intervention and the 2013 ACCF/AHA Guideline for the Management of ST-Elevation Myocardial Infarction. J Am Coll Cardiol. 2016 Mar 15;67(10):1235-1250. doi: 10.1016/j.jacc.2015.10.005. Epub 2015 Oct 21. No abstract available. PMID 26498666
- [Result] Engstrom T, Kelbaek H, Helqvist S, Hofsten DE, Klovgaard L, Holmvang L, Jorgensen E, Pedersen F, Saunamaki K, Clemmensen P, De Backer O, Ravkilde J, Tilsted HH, Villadsen AB, Aaroe J, Jensen SE, Raungaard B, Kober L; DANAMI-3-PRIMULTI Investigators. Complete revascularisation versus treatment of the culprit lesion only in patients with ST-segment elevation myocardial infarction and multivessel disease (DANAMI-3-PRIMULTI): an open-label, randomised controlled trial. Lancet. 2015 Aug 15;386(9994):665-71. doi: 10.1016/s0140-6736(15)60648-1. PMID 26347918